CLINICAL TRIAL: NCT06947226
Title: A Phase Ib/ll Clinical Study of Safety and Efficacy of 9MW2821 Monotherapy or Combined With Other Anticancer Therapy in Advanced Solid Tumors
Brief Title: A Clinical Study of 9MW2821 Monotherapy or Combined With Other Anticancer Therapy in Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9MW2821-CP201
Record Dates: First submitted 2025-04-21; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination Cohort (Experimental): Subjects will receive intravenous (IV) infusion of 9MW2821 + other anticancer therapy as per protocol
  Interventions: Drug: 9MW2821; Drug: Other anti-cancer therapy
- Single agent Cohort (Experimental): Subjects will receive intravenous (IV) infusion of 9MW2821 as per protocol
  Interventions: Drug: 9MW2821

INTERVENTIONS:
Drug: 9MW2821 — Subjects will receive intravenous (IV) infusion of 9MW2821 as per protocol
Drug: Other anti-cancer therapy — Subjects will receive other anticancer therapy as per protocol
  Arms: Combination Cohort

SUMMARY:
This study is a Phase Ib/ll, open-label, multicenter study designed to evaluate the safety and efficacy of 9MW2821 monotherapy or combined with other anticancer therapy in advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Competent to comprehend, sign, and date an independent ethics committee/institutional review board/research ethics board (IEC/IRB/REB) approved informed consent form.
2. Male or female subjects aged 18 to 75 years (including 18 and 75 years).
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Histopathological diagnosed of recurrent or locally advanced or metastatic solid tumors.
5. Adequate tumor tissues submitted for test.
6. Life expectancy of ≥ 12 weeks.
7. Subjects must have measurable disease according to RECIST (version 1.1).
8. Adequate organ functions.
9. Sexually active fertile subjects, and their partners, must agree to use contraception during the study and at least 6 months after termination of study therapy.
10. Subjects are willing to follow study procedures.

Exclusion Criteria:

1. History of another malignancy within 3 years before the first dose of study drug.
2. Ongoing clinically significant toxicities related to prior treatment.
3. Grade ≥ 2 peripheral neuropathy.
4. Severe or uncontrolled gastrointestinal diseases.
5. Other severe or uncontrolled diseases, including severe respiratory diseases, cardiovascular and cerebrovascular diseases of clinical significance.
6. Experienced clinically significant bleeding or had a clear bleeding tendency.
7. Central nervous system (CNS) metastasis and/or malignant meningitis.
8. Clinically significant pleural, abdominal, or pericardial effusion.
9. Chemotherapy or radiotherapy within 21 days prior to the first dose of study drug;
10. Known sensitivity to any of the ingredients of the investigational product; History of drug abuse or mental illness.
11. Pregnant and lactating women.
12. Other conditions that, in the Investigator's opinion, may not be suitable for the subject to be enrolled.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of AE/SAE (phase Ib) | Up to approximately 24 months
  Adverse event (AE), serious adverse event (SAE)
Objective Response Rate, ORR (phase II) | Up to approximately 24 months
  The proportion of participants with complete response (CR) or partial response (PR)

SECONDARY OUTCOMES:
Duration of Response, DOR | Up to approximately 24 months
  Time from the date of the first CR or PR to the earliest date of disease progression or death
Time To Response, TTR | Up to approximately 24 months
  Time from the date of first infusion to the date of CR or PR
Disease Control Rate, DCR | Up to approximately 24 months
  The percentage of subjects who experience CR, PR or stable disease (SD)
Progression-Free Survival, PFS | Up to approximately 24 months
  Time from the date of first infusion to the earliest date of disease progression or death
Overall Survival, OS | Up to approximately 24 months
  Time from the date of first infusion to the date of death
Pharmacokinetics parameter, Tmax | Up to approximately 24 months
  Peak time
Pharmacokinetics parameter, Cmax | Up to approximately 24 months
  Maximum concentration
Pharmacokinetics parameter, AUC | Up to approximately 24 months
  Area under the concentration-time curve
Pharmacokinetics parameter, t1/2 | Up to approximately 24 months
  Half-life
Pharmacokinetics parameter, V | Up to approximately 24 months
  Apparent volume of distribution
Pharmacokinetics parameter, CL | Up to approximately 24 months
  Clearance
Immunogenicity parameter | Up to approximately 24 months
  Anti-Drug Antibody (ADA) of 9MW2821

CONTACTS AND LOCATIONS:
Overall Officials: Feng Wang, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No